CLINICAL TRIAL: NCT00046774
Title: A Phase I, Open-Labeled, Dose-Ascending Clinical Trial of Immunotherapy of MRA, A Humanized Anti-IL 6 Receptor Monoclonal Antibody, In Patients With Systemic Lupus Erythematosus
Brief Title: Monoclonal Antibody Treatment for Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020272; 02-AR-0272
Record Dates: First submitted 2002-10-02; First posted 2002-10-03 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-09-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Safety; Nephritis; Biologic Therapy; Lymphocytes; Response; Lupus; Systemic Lupus Erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Nephritis

INTERVENTIONS:
Drug: MRA 003 US

SUMMARY:
This study will examine the safety and effects of the monoclonal antibody MRA in patients with systemic lupus erythematosus (SLE). Antibodies normally fight invading organisms. In autoimmune diseases, such as lupus, however, antibodies attack the body s own tissues. MRA is an antibody manufactured in the laboratory that blocks the action of interleukin-6 (IL-6), a substance that increases antibody production and is involved in inflammation that may cause organ damage in SLE.

Patients 18 years of age and older with moderately active systemic lupus erythematosus may be eligible for this 6-month study. Candidates will be screened with blood and urine tests, chest X-ray, electrocardiogram (EKG), and screening tests for certain cancers.

Participants will receive a total of up to seven infusions of MRA given every 2 weeks in the clinic. The MRA is infused over a period of about 1 hour through a catheter (thin plastic tube) inserted into an arm vein. Patients will be observed for 1 to 2 hours after each infusion for drug side effects. For the first and last infusions, patients will return to the clinic for blood tests 24 to 48 hours after the infusion. Additional tests may be done if medically indicated.

Three different doses of MRA will be used in three groups of patients. The first group (4 patients) will receive the lowest dose. If this dose is well tolerated, a second group (6 patients) will receive a higher dose. If this dose is also well tolerated, a third group (6 patients) will receive the highest study dose.

Patients will be evaluated at various intervals for up to 3 months after the last dose of MRA. The follow-up visits will include a review of the patient s medical history, a physical examination, blood and urine tests, and an EKG.

DETAILED DESCRIPTION:
Interleukin-6 (IL-6) levels are elevated in both human and murine systemic lupus erythematosus (SLE). Blocking the action of IL-6 ameliorates disease activity in murine models of SLE. MRA is a humanized monoclonal antibody against the human IL-6 receptor. Data from clinical trials in patients with rheumatoid arthritis suggest that MRA may be a safe agent to block the effect of IL-6 and therefore may be used to evaluate the effects of IL-6 blockade in patients with SLE. In this open label, dose-escalating, Phase I study, up to 27 subjects with moderately active SLE may be enrolled. Subjects will be treated with bi-weekly infusions of one of three doses (2mg/kg, 4 mg/kg or 8 mg/kg) of MRA for 12 weeks and followed for 8 weeks after the last dose. Patients with or without lupus nephritis may be enrolled if they do not require immediate immunosuppressive therapy other than prednisone at doses of less than or equal to 0.3 mg/kg/day. Safety will be evaluated using standard clinical and laboratory parameters. To assess the potential effect of MRA on SLE, clinical and laboratory evaluations and surrogate markers of inflammation and disease activity, such as autoantibody production and lymphocyte subsets, will be compared before and after the treatment. Patients who either do not tolerate the drug or those who have a clinically significant increase in their disease activity that does not respond to moderate doses of corticosteroids will be withdrawn from the protocol.

If this regimen is shown to be well tolerated, studies of efficacy will be planned. This agent is expected to be devoid of the most common toxicities of therapies commonly used in the treatment of SLE, such as myelosuppression, amenorrhea and osteoporosis.

This study will provide important preliminary information about the safety and possible effect of IL-6 blockade in SLE patients, an intervention that has been successful in animal models but has not yet been studied in humans.

ELIGIBILITY:
* IINCLUSION CRITERIA:

Age at entry at least 18 years

Must give written informed consent prior to entry in the protocol

Must fulfill at least 4 of the following criteria for SLE as defined by the American College of Rheumatology:

* Malar rash. Fixed Erythema, flat or raised, over the malar eminences.
* Discoid rash. Erythematous raised patches with adherent keratotic scaling and follicular plugging; atrophic scarring may occur.
* Photosensitivity. Exposure to UV light causes rash.
* Oral Ulcers. Includes oral and nasopharyngeal, observed by physician.
* Arthritis. Nonerosive arthritis involving two or more peripheral joints, characterized by tenderness, swelling or effusion.
* Serositis. Pleuritis or pericarditis documented by ECG or rub or evidence of pericardial effusion.
* Renal disorder. Proteinuria greater than 0.5 g/d or greater than 3+, or cellular casts.
* Neurologic disorder. Seizures without other cause or psychosis without other cause.
* Hematologic disorder. Hemolytic anemia or leukopenia (less than 4000/microL) or lymphopenia (less than 1500/microL) or thrombocytopenia (less than 100,000/microL) in the absence of offending drugs.
* Immunologic disorder. Anti-dsDNA, anti-Sm, and/or anti-phospholipid.
* Antinuclear antibodies. An abnormal titer of ANAs by immunofluorescence or an equivalent assay at any point in time in the absence of drugs known to induce ANAs.

Moderately active lupus not requiring immediate immunosuppressive therapy other than oral prednisone less than or equal to 0.3 mg/kg/day (or its equivalent). Moderately active lupus is defined by either of these two (a and b) sets of criteria:

a. Chronic glomerulonephritis with inadequate response to at least 6 months of adequate immunosuppressive therapy (with pulse methylprednisolone, cyclophosphamide, azathioprine, cyclosporine, mycophenolate mofetil or high dose daily corticosteroids, MTX or IV Ig), and

i. less than 30% increase in creatinine compared to lowest level during treatment,

ii. proteinuria less than or equal to 1.5 times the baseline before treatment,

iii. less than or equal to 2+ cellular casts in the urinary sediment (on a scale of 0-4), and

iv. Extra-renal disease activity does not exceed 10 on the non-renal components of the SELENA-SLEDAI score.

b. Patients with moderately active extra-renal lupus defined as an extra-renal SELENA-SLEDAI score in the range of 3 to 10, inclusive. The SELENA-SLEDAI score should have been stable for at least two weeks prior to screening.

One or more of the following:

i) Serum dsDNA level greater than or equal to 30 IU

ii) IgG anticardiolipin antibody levels greater than or equal to 20 GPL

iii) CRP greater than 0.8 mg/dL

iv) ESR greater than 25 mm/hr for men; ESR greater than 42 mm/hr for women.

Stable doses of prednisone less than or equal to 0.3 mg/kg/day (or its equivalent) for at least 2 weeks before the first treatment.

EXCLUSION CRITERIA:

Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening.

Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control during and for a period of three months after the completion of the study

Any therapy with human or murine antibodies or any experimental therapy within 3 months

Therapy with cyclophosphamide; pulse methylprednisolone or IV Ig within 4 weeks; or azathioprine, mycophenolate mofetil, cyclosporine or methotrexate within 2 weeks of first study treatment

Initiation or a change in the dose of an ACE-inhibitor within 2 weeks of first study treatment

Allergy to murine or human antibodies

History of anaphylaxis

Serum creatinine greater than 3.0 mg/dL

Active severe CNS lupus (encephalopathy, cerebrovascular accident, transverse myelitis, severe depression, psychosis)

Previous history of ischemic heart disease or evidence of ischemic heart disease on ECG

Congestive heart failure or cardiomyopathy

History of thrombosis or recurrent 2nd trimester abortions (3 or more) and elevated levels of anti-cardiolipin antibodies or lupus anticoagulant unless the patient is on anticoagulation

History of malignancy with the exception of basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix within the last 3 years

Active infection that requires the use of intravenous antibiotics and does not resolve within 1 week of Day 1

Any active viral infection that does not resolve within 10 days prior to Day 1

History of reactivation on EB viral infection or greater than 1,000 EBV genome equivalent/10(6) cells in PBMC preparations

Active hepatitis B, hepatitis C or HIV infection

WBC less than 3500/microL or ANC less than 3000/microL or Hgb less than 8.0 g/dL or platelets less than 50,000/microL or absolute lymphocyte count less than or equal to 500/microL.

ALT and/or AST greater than 2 times the upper limit of normal (ULN) or alkaline phosphatase greater than 1.5 times the ULN

Significant concurrent medical condition that, in the opinion of the principal investigator, could affect the patient's ability to tolerate or complete the study

Live vaccines within 4 weeks of first infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-09-02; Primary Completion 2007-01-01 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Safety/tolerance of MRA in pts w/SLE | Wks 0,2,6,12,14,20

SECONDARY OUTCOMES:
Clinical Pharmacokinetics of MRA | Wks 0,2,6,12,14,20

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kopf M, Baumann H, Freer G, Freudenberg M, Lamers M, Kishimoto T, Zinkernagel R, Bluethmann H, Kohler G. Impaired immune and acute-phase responses in interleukin-6-deficient mice. Nature. 1994 Mar 24;368(6469):339-42. doi: 10.1038/368339a0. PMID 8127368
- [Background] Bromander AK, Ekman L, Kopf M, Nedrud JG, Lycke NY. IL-6-deficient mice exhibit normal mucosal IgA responses to local immunizations and Helicobacter felis infection. J Immunol. 1996 Jun 1;156(11):4290-7. PMID 8666800
- [Background] Ramsay AJ, Husband AJ, Ramshaw IA, Bao S, Matthaei KI, Koehler G, Kopf M. The role of interleukin-6 in mucosal IgA antibody responses in vivo. Science. 1994 Apr 22;264(5158):561-3. doi: 10.1126/science.8160012.
- [Derived] Illei GG, Shirota Y, Yarboro CH, Daruwalla J, Tackey E, Takada K, Fleisher T, Balow JE, Lipsky PE. Tocilizumab in systemic lupus erythematosus: data on safety, preliminary efficacy, and impact on circulating plasma cells from an open-label phase I dosage-escalation study. Arthritis Rheum. 2010 Feb;62(2):542-52. doi: 10.1002/art.27221. PMID 20112381